CLINICAL TRIAL: NCT00901719
Title: Investigating the Interaction of Apelin and Systemic Angiotensin II Peripheral Resistance Vessels and Systemic Haemodynamics in Vivo in Man
Brief Title: Investigating Systemic and Local Vascular Responses to Apelin in the Context of Renin-angiotensin Upregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); British Heart Foundation (Other)
Responsible Party: Dr Gareth Barnes, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FS/09/019/26905 - 3
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2009-05

CONDITIONS: Heart Disease; Heart Failure; Vasodilatation
Keywords: Renin angiotensin system; Apelin; Cardiac output; Vasodilatation
MeSH Terms: conditions — Heart Diseases; Heart Failure; Aneurysm | interventions — Apelin; Acetylcholine; Nitroprusside

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium depletion (Experimental): Subjects will be randomised to normal diet or sodium depleted diet. The sodium depletion protocol comprises of a single oral dose of 40 mg of furosemide followed by an out-patient diet containing >2000 kcal of energy, >60 g of protein, <12 mmol of sodium and <70 mmol of potassium per day for 3 days prior to study. This diet is know to increase the activity of the renin-angiotensin system.
  Interventions: Drug: Apelin; Drug: Acetylcholine; Drug: Sodium nitroprusside; Drug: Systemic apelin infusion
- Normal diet (Placebo Comparator): Subjects will be randomised to a normal diet, with no restriction on sodium intake during the three days prior to the study.
  Interventions: Drug: Apelin; Drug: Acetylcholine; Drug: Sodium nitroprusside; Drug: Systemic apelin infusion

INTERVENTIONS:
Drug: Apelin — Using the technique of venous occlusive plethysmography subjects will receive three intrabrachial apelin infusions at 0.3, 1.0 and 3.0 nanomol/ml.
Drug: Acetylcholine — Using the technique of venous occlusive plethysmography subjects will receive three intrabrachial acetylcholine infusions at 5, 10 and 20 microg/min
Drug: Sodium nitroprusside — Using the technique of venous occlusive plethysmography subjects will receive three intrabrachial acetylcholine infusions at 1, 2 and 4 microg/min
Drug: Systemic apelin infusion — Following plethysmography patients will receive systemic infusion of (Pry)Apelin-13 (30, 100 and 300 nmol/min) for 5 mins cardiac output, blood pressure, heart rate and systemic vascular resistance will be measured at 5-min intervals.

SUMMARY:
The apelin-APJ system is a relatively new discovery. It has generated interest in part due to it's apparent ability to counteract the renin-angiotensin system, which is frequently overactive in many cardiovascular disease.

Two of the main actions of apelin are to increase the pumping ability of the heart and cause blood vessels to relax. The investigators wish to assess if these actions are altered in the setting of normal renin-angiotensin activation and increased renin-angiotensin activity.

ELIGIBILITY:
Inclusion Criteria:

* >18yr

Exclusion Criteria:

* Lack of informed consent
* Age < 18 years,
* Current involvement in other research studies,
* Systolic blood pressure >190 mmHg or <100 mmHg
* Malignant arrhythmias
* Renal or hepatic failure
* Haemodynamically significant aortic stenosis
* Severe or significant co morbidity
* Women of childbearing potential.
* Any regular medication
* Previous history of any cardiovascular disease

Ages: 18 Months to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output | 12 months
Change in apelin mediated vasodilatation | 12 months

SECONDARY OUTCOMES:
Change in systemic haemodynamics | 12 months
Change in relevant neurohumoral hormones | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Clincial Research Facility, Royal Infirmary of Edinburgh, 51 Little France Cresc, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Barnes GD, Alam S, Carter G, Pedersen CM, Lee KM, Hubbard TJ, Veitch S, Jeong H, White A, Cruden NL, Huson L, Japp AG, Newby DE. Sustained cardiovascular actions of APJ agonism during renin-angiotensin system activation and in patients with heart failure. Circ Heart Fail. 2013 May;6(3):482-91. doi: 10.1161/CIRCHEARTFAILURE.111.000077. Epub 2013 Mar 21. PMID 23519586